CLINICAL TRIAL: NCT01772771
Title: Molecular Testing for the MD Anderson Cancer Center Personalized Cancer Therapy Program
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA11-0852; NCI-2020-07334 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA11-0852 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-01-14; First posted 2013-01-21 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Melanoma; Sarcoma
MeSH Terms: conditions — Glioma; Hematologic Neoplasms; Melanoma; Sarcoma | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, saliva/buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection, chart review): Patients' previously collected tissue samples are analyzed. Patients may also undergo collection of blood, saliva or buccal samples for analysis. Patients' medical records are reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Testing; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, saliva/buccal swab samples
Other: Genetic Testing — Correlative studies
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Medical Chart Review — Review of medical records
  Other Names: Chart Review

SUMMARY:
This study performs standardized testing of tumor tissue samples to learn which genes are mutated (have changed) in order to provide personalized cancer therapy options to cancer patients at MD Anderson. This may help doctors use testing information on tumors to identify clinical trials that may be most relevant to patients. Researchers may also use the information learned from this study to develop a database of the different kinds of mutations in cancer-related genes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform molecular analysis for patients at MD Anderson to assist in personalized cancer therapy.

II. To determine the frequency of mutations, co-mutations and, other alterations including germline polymorphism and deleterious mutations (germline genetic factors), in cancer-related genes within different tumor types, and to determine patient preference for return of results.

III. To establish a database of somatic mutations, copy number alterations, gene fusion/translocation information and other biomarker alterations and clinical characteristics that can be used to select patients that may be eligible for new targeted therapy trials.

SECONDARY OBJECTIVES:

I. To determine enrollment to pathway-targeted therapy trials by cancer genotype and RNA and protein expression and plan additional pathway-targeted therapy trials.

II. To determine how somatic and/or germline mutations (including polymorphisms) in cancer-related genes, and other molecular alterations affect response to anti-tumor therapies and cancer outcomes and to determine how germline polymorphisms affect toxicity and side effects with cancer therapy.

III. To determine genomic alterations and other biomarkers detectable in plasma, exosomes or blood and their predictive value and evolution with treatment.

IV. To perform protein and RNA screening using different platforms such as immunohistochemistry (IHC), multiplex IHC, immunofluorescence (IF), mass spectrometry (MS), and Nanostring including assays from slides or tissue microarrays and image analysis strategies including digital pathology.

V. To determine feasibility of identifying actionable targets and rationale drug combinations based on gene expression profiling and systems biology.

VI. To determine feasibility of identifying novel antigens and other targets for novel strategies such as vaccines, immunotherapy and cell surface therapy.

VII. To use integrated biomarker and clinical data in conjunction with novel computational tools including large language models, machine learning, and other artificial intelligence tools for biomarker discovery and therapy-matching.

OUTLINE:

Patients' previously collected tissue samples are analyzed. Patients may also undergo collection of blood, saliva or buccal samples for analysis. Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically, radiographic, or cytologically documented cancer, suspected glioma, sarcoma, melanoma or hematologic cancer. Patients with benign tumors may also be consented at the discretion of the attending physician if molecular profiling is felt to have potential clinical implications.
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients may be consented without confirming the amount and quality of archival diagnostic or residual tissue available. However, research testing will only be performed on patients who have sufficient archived diagnostic tissue or residual tissue banked in one of the authorized tissue banks at MD Anderson available to proceed with testing. The extent of testing may be modified based on amount of tissue available. If any new tissue acquisition including a biopsy and/or surgical resection etc. is being ordered for clinical care or another research study, or an operation is being performed testing can be ordered on that sample
* Circulating cell-free deoxyribonucleic acid (cfDNA) Cohort: Circulating cell-free DNA next generation sequencing (NGS) testing will be performed with the Clinical Laboratory Improvement Act (CLIA)-certified Guardant360 panel (or equivalent) for select patients. This particular cohort of research collaboration will be supported by Guardant Health, Inc. at no charge to MD Anderson. Patients who are being considered for enrollment into clinical trials in the next 2 lines of therapy may be enrolled. Selected patients may have cfDNA, circulating RNA /exosome/circulating tumor cell testing approaches performed on alternate platforms (eg Foundation ACT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically, radiographic, or cytologically documented cancer, suspected glioma, sarcoma, melanoma or hematologic cancer
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2012-03-01 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of mutations and co-mutations | 20 years
  Will be assessed with descriptive statistics along with 95% Wilson score confidence intervals.
Distributions of mutations (including on gene expressions) | 20 years
  Distributions of mutations (including on gene expressions) between different tumor types and levels of clinical-pathological factors will be compared using the chi-squared test or Fisher's exact test, as appropriate for categorical variables
Database of somatic mutations and clinical characteristics | 20 years
  Collection and storage of tumor tissue specimens, blood and/or saliva samples of patients with cancer for somatic mutation analysis for assessing patients that may be eligible for new targeted therapy trials.

OTHER OUTCOMES:
Circulating cell free deoxyribonucleic acid (cfDNA) analysis | 20 years
  cfDNA analysis will be performed as an exploratory study to determine the concordance of specific alterations in the plasma and in tumor analysis, and to determine the change in cfDNA burden and mutation profile with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT01772771/ICF_000.pdf